CLINICAL TRIAL: NCT03952897
Title: Observational Study for the Assessment of Quality of Life Related to Health in Users of the Spa of Fitero (Navarra).
Brief Title: Quality of Life Related to Health in Spa Users
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Other Study IDs: EO-BALNEO-19
Record Dates: First submitted 2019-05-07; First posted 2019-05-16 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Knee Osteoarthritis; Hip Osteoarthritis; Rheumatoid Arthritis
Keywords: knee osteoarthritis; rheumatoid arthritis; balneology; hip balneology
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip; Arthritis, Rheumatoid | interventions — Balneology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Subjects treated with balneotherapy for 10 days, previously diagnosed with knee and/or hip osteoarthritis, and subjects previously diagnosed with rheumatoid arthritis.
  Interventions: Other: balneotherapy

INTERVENTIONS:
Other: balneotherapy — 10 days of balneotherapy with immersion techniques using Fitero spa water.

SUMMARY:
Hypothesis: The spa therapy treatment could improve health-related quality of life (HRQOL) in subjects with knee and/or hip osteoarthritis, and patients with rheumatoid arthritis.

Main objective: Analyze if HRQOL in patients with knee and/or hip osteoarthritis, and patients with rheumatoid arthritis is modified by spa therapy treatment in the spa of Fitero (Spain).

Design: Prospective observational study Participants: Fitero's spa users aged between 45-80 years old, diagnosed with knee and/or hip osteoarthritis, and also with rheumatoid arthritis. At least 40 patients of each type will be included in the study. Participants must be receiving a treatment of at least ten days.

Main Variable: The scores obtained in the Euroqol5Dimensions-5Levels questionnaire (EQ-5D-5L) (for all subjects), the Western Ontario MacMaster Universities Osteoarthritis Index (WOMAC) questionnaire, for subjects with knee and/or hip osteoarthritis, and the Health Assessment Questionnaire (HAQ), for subjects with rheumatoid arthritis.

Other variables: sociodemographic, anthropometric, clinics, and related with spa treatment.

Follow-up duration: 9 months.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed arthrosis of knee or hip and/or rheumatoid arthrosis
* balneotherapy treatment of at least 10 days.
* physically and mentally able to complete questionnaires

Exclusion Criteria:

* have followed a balneotherapy treatment in the six previous month

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Users of Fitero spa
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
HAQ (Health Assessment Questionnaire)-Disability of rheumatic patients | From 1st March 2019 to 1st December 2019
  Health Assessment Questionnaire (HAQ) assays the disability of rheumatic patients to carry out daily life activities. The questionary consists on 20 daily life questions, grouped in 8 areas, each one containing two or three questions related to daily life activities. Each question is scored from 0-3. 0 means "done without difficulties" (no disability), 3 score is "impossible to do" (completely disabled). The average of all responses is done. Average scores from 0-1 represent "mild to moderate difficulty", 1-2 means "moderate to severe disability", 3-2 indicates "severe to very severe disability".
WOMAC | From 1st March 2019 to 1st December 2019
  Western Ontario MacMaster Universities Osteoarthritis Index (WOMAC)

CONTACTS AND LOCATIONS:
Overall Officials: Inés Martínez-Galán, MD, Principal Investigator — University of Castilla-La Mancha
Locations (1):
- Universidad de Castilla-La Mancha, Toledo, Spain